CLINICAL TRIAL: NCT00521781
Title: Phase II Trial of Abraxane Plus Hormonal Therapy as Initial Treatment of Unresectable or Metastatic Adenocarcinoma of the Prostate
Brief Title: Study of Abraxane Plus Hormonal Therapy as Initial Treatment of Unresectable or Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMRI IRB#0407-0035; PCa-07-102 (Other: Principal Investigator)
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Unresectable or Metastatic Adenocarcinoma Prostate Cancer; Hormonal Therapy; Abraxane; M3thodist
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Albumin-Bound Paclitaxel; Leuprolide; Gonadotropin-Releasing Hormone; bicalutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment will be Abraxane/hormonal therapy (LHRH Agonist) for four nine-week cycles, followed by Total androgen blockade therapy (LHRH Agonist+ Anti-androgen) for 2 years from the time the hormonal therapy was started.
  Interventions: Drug: Abraxane; Drug: Leuprolide; Drug: Bicalutamide

INTERVENTIONS:
Drug: Abraxane — 100 mg/m2 IVPB Day 1, 8, 15, 22, 29,36,43,50 of each cycle for 4 nine-week cycles (Each cycle of Abraxane/hormonal therapy will consist of 8 weeks of Abraxane therapy and 1 week of rest.)
Drug: Leuprolide — 7.5 mg monthly or 22.5 mg quarterly, can begin within 3 months of initiating Abraxane for 2 years
  Other Names: Depot Lupron®; LHRH agonist
Drug: Bicalutamide — 50 mg p.o. daily starts week 36 of initiating Abraxane.
  Other Names: Casodex®; Anti-androgen therapy

SUMMARY:
The purpose of the clinical trial is to assess the clinical benefit as measured by time to tumor progression of Abraxane plus hormonal therapy when applied to previously untreated patients with unresectable or metastatic adenocarcinoma of the prostate, as well as to assess safety and tolerability of the study drug regimen and to evaluate secondary efficacy endpoints such as overall survival and duration of response.

DETAILED DESCRIPTION:
Abraxane is a potent anticancer drug that stops cancer cells from growing and dividing by interfering with certain cell structures and killing the cancer cells. Abraxane is the first albumin-bound taxane particle of approximately 130 nanometers that takes advantage of albumin, a natural carrier of water-insoluble molecules (e.g., various nutrients, vitamins, and hormones) found in humans. Albumin is a protein that acts as the body's key transporter of nutrients and other water-insoluble molecules and selectively accumulates in tumor tissues.

The delivery of chemotherapy/hormone therapy in a setting of androgen-independent prostate cancer has demonstrated: survival benefit associated with a PSA decline and tolerable toxicity, thus strongly suggesting that disease modifying potential exists. Preclinical data supports the benefit of simultaneous chemotherapy/hormonal therapy and androgen deprivation. The stage is set for chemotherapy/hormonal therapy to be given earlier in men with prostate cancer. Data suggests a transformation from an androgen-dependent to an androgen-independent phenotype is mediated by the expansion of an androgen-independent clone already present at the time of androgen deprivation. If this model is correct, it would be feasible to bring chemotherapy/hormonal therapy up front when the corresponding tumor burden is minimal.

It is hoped that by bringing therapy against all components of the tumor initially, the emergence of androgen-independent growth will be delayed, ultimately prolonging patient survival. This study will test this hypothesis of Abraxane plus hormonal therapy followed by standard hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of adenocarcinoma of the prostate.
* Patients must belong to one of four groups: 1) Local/Regional with prior definitive therapy: Patients with local/regional recurrence following prostatectomy or radiation therapy who still have a normal bone scan. 2) Local/Regional without prior definitive therapy: Patients felt to be unresectable, or are felt not to be candidates for, radiation therapy. 3) Low volume bone disease: Patients with 1 or 2 bone metastases. 4) High volume bone/visceral disease: Patients with ≥ 3 metastatic bone sites or visceral metastases.
* Patients meeting these criteria are eligible even without any radiographically demonstrable abnormality. All patients must have an elevated PSA prior to initial hormone exposure defined as: 1) For patients with prior prostatectomy, the PSA must be rising with an associated doubling time of ≤ 3 months. 2) For patients with prior radiation therapy, the PSA must be ≥ 1.0 ng/mL with an associated doubling time of ≤ 3 months. 3) For patients with the prostate in place, the PSA must be elevated with biopsy proven disease and are not candidates for local therapy.
* Patients may be on an LHRH agonist (with or without an anti-androgen), or already medically castrated, at the time of study entry, provided such therapy was started within 3 months of study entry.
* No previous cytotoxic systemic therapy of any kind is allowed, including systemic irradiation with strontium-89 and samarium. Previous definitive radiotherapy to one metastatic site is acceptable. At least 8 weeks must have elapsed since radiation therapy to the pelvis. Patients having limited irradiation of a single metastatic site are eligible 4 weeks following the completion of radiation.
* Patients may have had previous exposure to androgen deprivation therapy if it was given for ≤ 6 months to, "downstage" the primary, and provided such therapy completed at least 12 months prior to entry into this study.
* Patients must be free of serious co-morbidity and have a life expectancy of ≥ 3 years.
* Patients must have adequate physiologic reserves as evidenced by Zubrod Performance Status (ZPS) of ≤ 2, adequate bone marrow function, renal function and liver function and no evidence of active ischemia on ECG (if clinically indicated, documentation of EF ≥ 40%.)

Exclusion Criteria:

* Patients must not have a second malignancy unless there is confidence of previous curative therapy.
* Patients with a recent history of TIA (within 6 months), or are requiring regular antianginal therapy or are having claudication sufficient to limit activity are not eligible. Patients with a previous history of deep venous thrombosis or pulmonary embolism (within 12 months) are not eligible.
* Patients must not have a serious intercurrent medical or psychiatric illness, including serious active infection.
* Patients must not have Sensory neuropathy of grade 1 or greater.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Assess the clinical benefit as measured by time to tumor progression of Abraxane plus hormonal therapy when applied to previously untreated patients with unresectable or metastatic adenocarcinoma of the prostate. | measurements every 4 wks while on Abraxane; then every 12 wks

SECONDARY OUTCOMES:
Assess safety and tolerability of the study drug regimen. Overall survival Duration of response PSA "lead-time" to symptomatic or radiographic progression. | AEs as occur

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Baylor College of Medicine - Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No